CLINICAL TRIAL: NCT01700192
Title: A One-year Placebo-Controlled Study Evaluating the Efficacy and Safety of the House Dust Mite Sublingual Allergen Immunotherapy Tablet (SCH 900237/MK 8237) in Children and Adult Subjects With House Dust Mite-Induced Allergic Rhinitis/Rhinoconjunctivitis With or Without Asthma (Protocol No. P05607/001)
Brief Title: Efficacy and Safety Study of SCH 900237/MK-8237 in Children and Adults With House Dust Mite-Induced Allergic Rhinitis/Rhinoconjunctivitis (P05607)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: ALK-Abelló A/S (Industry)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: P05607; MK-8237-001 (Other: Merck Protocol ID)
Record Dates: First submitted 2012-10-02; First posted 2012-10-04 (Estimated); Results first posted 2017-03-03 (Actual); Last update posted 2017-09-15 (Actual); Status verified 2017-09

CONDITIONS: Rhinitis, Allergic, Perennial; Rhinitis, Allergic, Nonseasonal
MeSH Terms: conditions — Rhinitis, Allergic, Perennial

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- MK-8237 (Experimental): MK-8237 12 Development Units (DU) rapidly dissolving tablets administered sublingually once daily (q.d.).
  Interventions: Biological: MK-8237 tablets; Drug: Rescue Medication: Self-Injectable Epinephrine; Drug: Rescue Medication: Loratadine tablets; Drug: Rescue Medication: Olopatadine ophthalmic drops; Drug: Rescue Medication: Mometasone furoate nasal spray
- Placebo (Placebo Comparator): Placebo to MK-8237 rapidly dissolving tablets administered sublingually q.d.
  Interventions: Biological: Placebo tablets; Drug: Rescue Medication: Self-Injectable Epinephrine; Drug: Rescue Medication: Loratadine tablets; Drug: Rescue Medication: Olopatadine ophthalmic drops; Drug: Rescue Medication: Mometasone furoate nasal spray

INTERVENTIONS:
Biological: MK-8237 tablets — MK-8237 12 DU rapidly dissolving tablets administered sublingually q.d.
  Other Names: SCH 900237
  Arms: MK-8237
Biological: Placebo tablets — Placebo to MK-8237 rapidly dissolving tablets administered sublingually q.d.
  Arms: Placebo
Drug: Rescue Medication: Self-Injectable Epinephrine — Self-injectable epinephrine (preferred dose of 0.30 mg) administered intramuscularly as needed for rescue medication.
Drug: Rescue Medication: Loratadine tablets — Loratadine tablet 10 mg administered orally as needed for rescue medication.
Drug: Rescue Medication: Olopatadine ophthalmic drops — Olopatadine hydrochloride ophthalmic drops 0.1% administered as needed for rescue medication.
Drug: Rescue Medication: Mometasone furoate nasal spray — Mometasone furoate monohydrate nasal spray 50 mcg administered intranasally as needed for rescue medication.

SUMMARY:
The purpose of this study is to assess the efficacy and safety of MK-8237 (SCH 900237) in the treatment of House Dust Mite (HDM)-Induced Allergic Rhinitis/Rhinoconjunctivitis (AR/ARC) in children and adults.

The primary hypothesis of this study is that administration of MK-8237, compared to placebo, results in significant reduction in the average total combined rhinitis score (TCRS).

ELIGIBILITY:
Inclusion Criteria:

* History of AR/ARC to house dust of 1 year duration or more (with or without asthma)
* If female of childbearing potential, has a negative urine pregnancy test at Screening and agrees to remain abstinent or use (or have their partner use) an acceptable method of birth control within the projected duration of the study
* Able to read, understand and complete questionnaires and diaries

Exclusion Criteria:

* Clinically relevant history of symptomatic ARC caused by animal dander, molds and/or cockroach (e.g. present in the home, job, daycare, etc.) or other perennial allergen
* History of symptomatic seasonal ARC and/or asthma due to an allergen to which the participant is sensitized and regularly exposed
* Nasal condition that could confound the efficacy or safety assessments (e.g., nasal polyposis)
* Received an immunosuppressive treatment within 3 months prior to screening
* Unstable or severe asthma, or has experienced a life-threatening asthma attack or an occurrence of any clinical deterioration of asthma that resulted in emergency treatment, hospitalization due to asthma, or treatment with systemic corticosteroids (but allowing short-acting beta agonists [SABAs]) at any time within 3 months prior to screening
* Asthma requiring high-dose inhaled corticosteroids (ICS) within 6 months prior to screening
* History of anaphylaxis with cardiorespiratory symptoms with prior immunotherapy, unknown cause or inhalant allergen
* History of chronic urticaria and/or angioedema within 2 years prior to screening
* History of chronic sinusitis during 2 years prior to screening
* Pregnant, breastfeeding, or expecting to conceive within the projected duration of the study
* Previous immunotherapy treatment with any HDM allergen for more than 1 month within 5 years prior to screening
* Previous exposure to MK-8237
* Receiving ongoing treatment with any specific immunotherapy at screening
* Known history of allergy, hypersensitivity or intolerance to investigational medicinal products (except for D. pteronyssinus and/or D. farinae), rescue medications or self-injectable epinephrine
* Unable to meet medication washout requirements prior to screening
* Unable or unwilling to comply with the use of self-injectable epinephrine
* Business or personal relationship with investigational site personnel or Sponsor who is directly involved with the conduct of the study
* Likely to travel for extended periods of time during the efficacy assessment period
* Participating in a different investigational study at any site during this study

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1482 (Actual)
Dates: Start 2013-01; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

REFERENCES:
- [Result] Nolte H, Bernstein DI, Nelson HS, Kleine-Tebbe J, Sussman GL, Seitzberg D, Rehm D, Kaur A, Li Z, Lu S. Efficacy of house dust mite sublingual immunotherapy tablet in North American adolescents and adults in a randomized, placebo-controlled trial. J Allergy Clin Immunol. 2016 Dec;138(6):1631-1638. doi: 10.1016/j.jaci.2016.06.044. Epub 2016 Aug 10. PMID 27521719
- [Derived] Horn A, Bernstein DI, Okubo K, Dalgaard T, Hels O, Sorensen HF, Henriksen M, Azuma R, Mikler J, Nolte H. House dust mite sublingual immunotherapy tablet safety in adolescents with allergic rhinoconjunctivitis: Worldwide clinical trial results. Ann Allergy Asthma Immunol. 2023 Jun;130(6):797-804.e2. doi: 10.1016/j.anai.2023.03.006. Epub 2023 Mar 15. PMID 36924936
- [Derived] Fortescue R, Kew KM, Leung MST. Sublingual immunotherapy for asthma. Cochrane Database Syst Rev. 2020 Sep 14;9(9):CD011293. doi: 10.1002/14651858.CD011293.pub3. PMID 32926419
- [Derived] Bernstein DI, Kleine-Tebbe J, Nelson HS, Bardelas JA Jr, Sussman GL, Lu S, Rehm D, Svanholm Fogh B, Nolte H. SQ house dust mite sublingual immunotherapy tablet subgroup efficacy and local application site reaction duration. Ann Allergy Asthma Immunol. 2018 Jul;121(1):105-110. doi: 10.1016/j.anai.2018.04.007. Epub 2018 Apr 12. PMID 29656145
- [Derived] Nolte H, Bernstein DI, Sussman GL, Svanholm Fogh B, Lu S, Husoy B, Nelson HS. Impact of Adverse Event Solicitation on the Safety Profile of SQ House Dust Mite Sublingual Immunotherapy Tablet. J Allergy Clin Immunol Pract. 2018 Nov-Dec;6(6):2081-2086.e1. doi: 10.1016/j.jaip.2018.01.037. Epub 2018 Feb 10. PMID 29432959

RESULTS

PARTICIPANT FLOW:
Groups:
- MK-8237: Participants took MK-8237 12 development unit (DU) rapidly dissolving tablets administered sublingually once daily (q.d.) for up to one year.
- Placebo: Participants took placebo to MK-8237 rapidly dissolving tablets administered sublingually q.d. for up to one year.
Period: Overall Study
Arm/Group | MK-8237 | Placebo
Started | 741 | 741
Treated | 740 | 741
All Participants as Treated (APaT) | 743 (Three participants randomized to receive placebo were given MK-8237 12 DU.) | 738 (Three participants randomized to receive placebo were given MK-8237 12 DU.)
Completed | 561 | 613
Not Completed | 180 | 128
Not completed — Adverse Event | 73 | 18
Not completed — Lack of Efficacy | 1 | 0
Not completed — Lost to Follow-up | 42 | 29
Not completed — Noncompliance with study drug | 0 | 5
Not completed — Physician Decision | 2 | 3
Not completed — Pregnancy | 1 | 4
Not completed — Progressive disease | 1 | 0
Not completed — Protocol Violation | 3 | 4
Not completed — Technical problems | 0 | 1
Not completed — Withdrawal by Subject | 56 | 64
Not completed — Never received study drug | 1 | 0

BASELINE CHARACTERISTICS:
Population: Baseline Characteristics refer to all randomized participants.
Groups:
- MK-8237: Participants took MK-8237 12 DU rapidly dissolving tablets administered sublingually q.d. for up to one year.
- Total: Total of all reporting groups
Arm/Group | MK-8237 | Placebo | Total
Number analyzed (Participants) | 741 | 741 | 1482
Age, Continuous [Mean (Standard Deviation); unit: Years] | 34.9 (13.82) [12 to 77] | 35.2 (13.74) [12 to 85] | 35.1 (13.77) [12 to 85]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 445 | 430 | 875
  Male | 296 | 311 | 607

OUTCOME MEASURES:

1. Primary Outcome: Average Total Combined Rhinitis Score (TCRS) During Last 8 Weeks of Treatment
Description: The TCRS is the sum of the rhinitis Daily Symptom Score (DSS; range: 0 to 12) and the rhinitis Daily Medication Score (DMS; range: 0 to 12); the total possible TCRS ranges from 0 to 24 points with higher scores indicative of greater symptom severity. The endpoint was calculated as the average daily diary entry score from the last 8 weeks of treatment.
Time Frame: Last 8 weeks of treatment (Weeks 44 to 52)
Population: The analysis population consists of all randomized participants who received at least 1 dose of study drug and had data available.
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | MK-8237 | Placebo
Number analyzed (Participants) | 566 | 620
Score on a Scale | 4.67 (3.55) | 5.49 (3.82)
Statistical Analysis 1: Comparison: MK-8237 vs Placebo; Test type: Superiority or Other; p < 0.001, Wilcoxon (Mann-Whitney); Median Difference (Final Values) = -0.80, 95% CI 2-sided [-1.20 to -0.40]
Statistical Analysis 2: Comparison: MK-8237 vs Placebo; Test type: Superiority or Other; Treatment Difference Relative to Placebo = -17.2, 95% CI 2-sided [-25.0 to -9.7]

2. Primary Outcome: Number of Participants Who Experience At Least One Adverse Event (AE)
Description: An AE is defined as any untoward medical occurrence in a clinical investigation participant administered a pharmaceutical product and which does not necessarily have to have a causal relationship with this treatment.
Time Frame: Up to 54 weeks
Population: The All Participants as Treated (APaT) population consists of all randomized participants who received at least 1 dose of study drug (data presented according to actual treatment received).
Measure: Number; unit: Participants
Arm/Group | MK-8237 | Placebo
Number analyzed (Participants) | 743 | 738
Participants | 676 | 539

3. Primary Outcome: Number of Participants Who Discontinue Study Drug Due to an AE
Description: as for outcome 2
Time Frame: Up to 52 weeks
Population: The APaT population consists of all randomized participants who received at least 1 dose of study drug (data presented according to actual treatment received).
Measure: Number; unit: Participants
Arm/Group | MK-8237 | Placebo
Number analyzed (Participants) | 743 | 738
Participants | 73 | 19

4. Secondary Outcome: Average Rhinitis Daily Symptom Score (Rhinitis DSS) During Last 8 Weeks of Treatment
Description: The Rhinitis DSS ranges from a score of 0 to 12 (higher scores indicative of greater symptom severity). The endpoint was calculated as the average daily diary entry score from the last 8 weeks of treatment.
Time Frame: Last 8 weeks of treatment (Weeks 44 to 52)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | MK-8237 | Placebo
Number analyzed (Participants) | 566 | 620
Score on a Scale | 3.83 (2.64) | 4.46 (2.80)
Statistical Analysis 1: Comparison: MK-8237 vs Placebo; Test type: Superiority or Other; p < 0.001, Wilcoxon (Mann-Whitney); Median Difference (Final Values) = -0.60, 95% CI 2-sided [-1.00 to -0.30]
Statistical Analysis 2: Comparison: MK-8237 vs Placebo; Test type: Superiority or Other; Treatment Difference Relative to Placebo = -15.5, 95% CI 2-sided [-24.4 to -7.3]

5. Secondary Outcome: Average Rhinitis Daily Medication Score (Rhinitis DMS) During Last 8 Weeks of Treatment
Description: The Rhinitis DMS ranges from a score of 0 to 12 (higher scores indicative of greater symptomatic medication use). The endpoint was calculated as the average daily diary entry score from the last 8 weeks of treatment.
Time Frame: Last 8 weeks of treatment (Weeks 44 to 52)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | MK-8237 | Placebo
Number analyzed (Participants) | 566 | 620
Score on a Scale | 0.84 (1.817) | 1.03 (2.074)
Statistical Analysis 1: Comparison: MK-8237 vs Placebo; Test type: Superiority or Other; p = 0.154, Zero-inflated Log-normal Model; Mean Difference (Final Values) = -0.15, 95% CI 2-sided [-0.35 to 0.05]
Statistical Analysis 2: Comparison: MK-8237 vs Placebo; Test type: Superiority or Other; Treatment Difference Relative to Placebo = -18.4, 95% CI 2-sided [-41 to 4.3]

6. Secondary Outcome: Average Total Combined Rhinoconjunctivitis Score (TCS) During Last 8 Weeks of Treatment
Description: The TCS is the sum of the rhinoconjunctivitis DSS (rhinitis DSS and conjunctivitis DSS; range: 0 to 18) and the rhinoconjunctivitis DMS (rhinitis DMS and conjunctivitis DMS; range: 0 to 20); the total possible TCS ranges from 0 to 38 points with higher scores indicative of greater symptom severity. The endpoint was calculated as the average daily diary entry score from the last 8 weeks of treatment.
Time Frame: Last 8 weeks of treatment (Weeks 44 to 52)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | MK-8237 | Placebo
Number analyzed (Participants) | 566 | 620
Score on a Scale | 6.40 (5.16) | 7.62 (5.48)
Statistical Analysis 1: Comparison: MK-8237 vs Placebo; Test type: Superiority or Other; p < 0.001, Wilcoxon (Mann-Whitney); Median Difference (Final Values) = -1.10, 95% CI 2-sided [-1.70 to -0.60]
Statistical Analysis 2: Comparison: MK-8237 vs Placebo; Test type: Superiority or Other; Treatment Difference Relative to Placebo = -16.7, 95% CI 2-sided [-24.6 to -4.0]

7. Secondary Outcome: Average Allergic Rhinitis/Rhinoconjunctivitis Symptoms Assessed by Visual Analogue Scale (VAS) During Last 8 Weeks of Treatment
Description: Participants indicated the severity of symptoms in the past week on a VAS with a score range of 0 ("no symptoms") to 100 ("severe symptoms"). Symptoms were assessed during 2 clinic visits occurring during the final 8 weeks of treatment (VAS score reflects the mean of 2 scores).
Time Frame: Last 8 weeks of treatment (Weeks 44 to 52)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | MK-8237 | Placebo
Number analyzed (Participants) | 540 | 585
Score on a Scale | 42.29 (23.57) | 47.96 (23.66)
Statistical Analysis 1: Comparison: MK-8237 vs Placebo; Test type: Superiority or Other; p < 0.001, Wilcoxon (Mann-Whitney); Median Difference (Final Values) = -6.10, 95% CI 2-sided [-9.10 to -3.10]
Statistical Analysis 2: Comparison: MK-8237 vs Placebo; Test type: Superiority or Other; Treatment Difference Relative to Placebo = -16.0, 95% CI 2-sided [-22.7 to -8.3]

ADVERSE EVENTS:
Time Frame: Up to 54 weeks
Description: The APaT population consists of all randomized participants who received at least 1 dose of study drug (data presented according to actual treatment received).
Groups:
- MK-8237 12 DU: Participants took MK-8237 12 DU rapidly dissolving tablets administered sublingually q.d. for up to one year.
Arm/Group | MK-8237 12 DU | Placebo
Serious Adverse Events (participants affected / at risk) | 11/743 | 7/738
Other Adverse Events (participants affected / at risk) | 642/743 | 389/738
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MK-8237 12 DU (N=743) | Placebo (N=738)
Pericarditis (Cardiac disorders) | 1 (1) | 0 (0)
Tympanic membrane perforation (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Oral pain (Gastrointestinal disorders) | 1 (1) | 0 (0) — Due to overdose; classified as SAE by sponsor but does not meet International Council for Harmonisation (ICH) SAE criteria.
Oral pruritus (Gastrointestinal disorders) | 1 (1) | 0 (0) — Due to overdose; classified as SAE by sponsor but does not meet ICH SAE criteria.
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Anaphylactic reaction (Immune system disorders) | 0 (0) | 1 (1)
Food allergy (Immune system disorders) | 0 (0) | 1 (1)
Diverticulitis (Infections and infestations) | 1 (1) | 0 (0)
Infected bites (Infections and infestations) | 1 (1) | 0 (0)
Peritonitis (Infections and infestations) | 1 (1) | 0 (0)
Concussion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Hepatic cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0)
Bipolar I disorder (Psychiatric disorders) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 0 (0) | 1 (1)
Calculus ureteric (Renal and urinary disorders) | 1 (1) | 0 (0)
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) — Due to overdose; classified as SAE by sponsor but does not meet ICH SAE criteria.
Deep vein thrombosis (Vascular disorders) | 1 (1) | 0 (0)
Hypertensive emergency (Vascular disorders) | 1 (1) | 0 (0)
Alcohol abuse (Psychiatric disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MK-8237 12 DU (N=743) | Placebo (N=738)
Ear pruritus (Ear and labyrinth disorders) | 382 (1637) | 92 (244)
Abdominal pain upper (Gastrointestinal disorders) | 92 (212) | 44 (87)
Diarrhoea (Gastrointestinal disorders) | 55 (85) | 27 (42)
Glossodynia (Gastrointestinal disorders) | 119 (296) | 26 (58)
Lip swelling (Gastrointestinal disorders) | 140 (353) | 19 (42)
Mouth swelling (Gastrointestinal disorders) | 73 (165) | 12 (32)
Mouth ulceration (Gastrointestinal disorders) | 85 (196) | 27 (41)
Nausea (Gastrointestinal disorders) | 121 (293) | 57 (111)
Oral pruritus (Gastrointestinal disorders) | 468 (1966) | 109 (277)
Palatal swelling (Gastrointestinal disorders) | 82 (183) | 11 (14)
Paraesthesia oral (Gastrointestinal disorders) | 71 (173) | 21 (28)
Swollen tongue (Gastrointestinal disorders) | 123 (255) | 17 (31)
Tongue ulceration (Gastrointestinal disorders) | 96 (232) | 21 (29)
Nasopharyngitis (Infections and infestations) | 62 (81) | 61 (68)
Upper respiratory tract infection (Infections and infestations) | 63 (76) | 74 (87)
Dysgeusia (Nervous system disorders) | 73 (143) | 29 (48)
Headache (Nervous system disorders) | 35 (43) | 47 (63)
Pharyngeal oedema (Respiratory, thoracic and mediastinal disorders) | 109 (268) | 23 (40)
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 506 (2144) | 172 (505)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor must have the opportunity to review all proposed abstracts, manuscripts or presentations regarding this trial 45 days prior to submission for publication/presentation.